CLINICAL TRIAL: NCT02366559
Title: Comparing the Efficacy and Risk of Adverse Events of Electrocautery Versus 532 nm Qswitched Neodymium-doped Yttrium Aluminium Garnet Laser for the Treatment of Flat Seborrheic Keratoses: A Randomized Control Trial
Brief Title: Electrocautery vs Q-switch for Seborrheic Keratosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU105340
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Keratosis, Seborrheic
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electrocautery (Active Comparator): Blocks of subjects' lesions will be randomized 1:1 to receive electrocautery or 532 nm Nd:YAG laser. Prior to treatment with either electrocautery or 532nm Q-switched Nd:YAG laser, a topical EMLA cream will be applied to the lesions for at least 60 minutes under occlusion at the area of treatment.
  Interventions: Device: Hyfrecator
- 532 nm Nd:YAG laser (Active Comparator): Blocks of subjects' lesions will be randomized 1:1 to receive electrocautery or 532 nm Nd:YAG laser. Prior to treatment with either electrocautery or 532nm Q-switched Nd:YAG laser, a topical EMLA cream will be applied to the lesions for at least 60 minutes under occlusion at the area of treatment.
  Interventions: Device: 532 nm Q-switched Nd:YAG laser

INTERVENTIONS:
Device: Hyfrecator
  Arms: electrocautery
Device: 532 nm Q-switched Nd:YAG laser
  Arms: 532 nm Nd:YAG laser

SUMMARY:
The primary objective of this study is to compare the efficacy and risk of adverse events of electrocautery versus 532 nm Q-switched neodymium-doped yttrium aluminium garnet (Nd:YAG) laser for the treatment of flat seborrheic keratoses.

This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are Caucasian or Asian.
2. Subjects who are between 18-65 year olds.
3. Subjects have flat or macular seborrheic keratosis on dorsum of the hands and wrists, extensor surfaces of the forearms. The diagnosis of flat seborrheic keratosis is confirmed by two clinical dermatologists using routine clinical examination and dermoscopy.
4. Subjects have Fitzpatrick skin type I-III.
5. Subjects are in good health.
6. Subjects have the willingness and the ability to understand and provide informed consent and communicate with the investigator.

Exclusion Criteria:

1. History of keloids or hypertrophic scars.
2. Pregnant or lactating or intends to become pregnant in the next 3 months.
3. Active skin disease or skin infection in the treatment area.
4. Previous history of lidocaine allergy.
5. History of methemoglobinemia
6. Unable to understand the protocol or to give informed consent.
7. Any other condition that would, in the professional opinion of the investigator, potentially affect response or participation in the clinical study or would pose as an unacceptable risk to subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pigmentation from baseline to week 18 | Baseline and 18 weeks
  Blinded photo raters will the lesion pigmentation on a scale of -50 (most hypopigmented relative to baseline) to +50 (most hyperpigmented relative to baseline) for both treatments.
Change in lesion texture from baseline to week 18 | Baseline and 18 weeks
  Blinded photo raters will the lesion texture on a scale of -50 (most worsening relative to baseline) to +50 (most improvement relative to baseline) for both treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University